CLINICAL TRIAL: NCT06296654
Title: Effect of Empowerment-Based Interventions on Self-Efficacy and Self-Care Capacity Among Adults With Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bahrain (Other)
Responsible Party: Principal Investigator, Zohour Ibrahim Mahmoud Rashwan, Assistant Professor, University of Bahrain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 25/2021-22 dt. Dec. 12,2021
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Self-Efficacy; Self-Care
Keywords: Sickle Cell Disease; Self-efficacy; Self-Management; Activities of Daily Living
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empowerment-Based Interventions (EBI) (Experimental): The EBI was used for the study group. It is an integrative educational program under the patient-centered care approach emphasizing collaborative patient interaction. The EBI was implemented through structured (a) small-group discussion sessions, (b) individualized consultations, and (c) follow-up sessions.
  Interventions: Behavioral: Empowerment-Based Interventions
- standard health education (Active Comparator): Patients in the control group received standard health education from SCD clinics in the HC. The clinic employs a multidisciplinary team, including a nurse, a physician, a health record clerk, a laboratory technician, a social worker, and a health promotion specialist, to provide integrated patient health services. It consists of both preventative and curative services. The nurses at the health center provide patients with information regarding factors that may cause vaso-occlusion and precipitate VOCs when to seek emergency care and educate patients on the significance of regular medical examinations and screening using different standardized audiovisual aids.
  Interventions: Behavioral: Standard Health Education

INTERVENTIONS:
Behavioral: Empowerment-Based Interventions — The Empowerment-Based Interventions was used for the study group. It is an integrative educational program under the patient-centered care approach emphasizing collaborative patient interaction. The EBI was implemented through structured (a) small-group d
  Arms: Empowerment-Based Interventions (EBI)
Behavioral: Standard Health Education — Patients in the control group received standard health education from SCD clinics in the HC. The clinic employs a multidisciplinary team, including a nurse, a physician, a health record clerk, a laboratory technician, a social worker, and a health promotion specialist, to provide integrated patient health services. It consists of both preventative and curative services. The nurses at the health center provide patients with information regarding factors that may cause vaso-occlusion and precipitate VOCs when to seek emergency care and educate patients on the significance of regular medical examinations and screening using different standardized audiovisual aids.
  Arms: standard health education

SUMMARY:
This study aimed to To investigate the effect of empowerment-based interventions (EBI) on self-efficacy and self-care capacity among adults with Sickle Cell Disease (SCD).

The hypotheses of this study were: Adults with SCD who receive EBI exhibit higher self-efficacy, self- management capacity and HRQoL than those who do not.

DETAILED DESCRIPTION:
A pre-test-post-test control group experimental study was conducted at two randomly selected health centers in Bahrain using a cluster sampling technique. A sample of 68 out of 122 adults with SCD was randomly assigned to two groups. The EBI was implemented through structured small-group discussion sessions, individualized consultations, and follow-up sessions. Individualized consultations for self-management were done by adopting the 5A model (assess, advise, agree, assist, and arrange). Weekly communication was done to check the patient's progress, and both groups were re-evaluated for self-efficacy and self-care capacity after one month.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with SCD f
* Receiving treatment from primary health care facilities
* Able to read and write
* Having the chance to attend the educational sessions .

Exclusion Criteria:

* A history of mental illness .

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-22 (Actual)

PRIMARY OUTCOMES:
Sickle Cell Self-Efficacy | 1 month
  This scale was designed by Edwards et al. (2000) to assess the self-appraisals of adult patients with sickle cell disease for their ability to engage in daily functional activities(22). It is composed of nine items rated on a five-point Likert scale ranging from "not at all sure" to "very sure cell disease for their ability to engage in daily functional activities. It is composed of nine items rated on a five-point Likert scale ranging from "not at all sure" to "very sure." The total score ranged from 9 to 45, with higher scores indicating higher levels of self-efficacy.

SECONDARY OUTCOMES:
Self-Care Capacity | 1 month
  This scale was originally developed by Kearney and Fleischer (1979) according to Orem's self-care theory and revised by Wang and Laffrey (2000) to assess the level of health-related self-care capacity(24,25). The scale consists of 15 items, rated on a 5-point Likert scale ranging from "totally disagree" (1 point) to "totally agree" (5 points).

CONTACTS AND LOCATIONS:
Overall Officials: adnan Bekhit, Professor, Study Chair — College of Health and Sport Sciences, University of Bahrain
Locations (1):
- College of Health and Sport Sciences, University of Bahrain, Manama, Bahrain

REFERENCES:
- [Background] Al Raqaishi H, Al Qadire M, Alzaabi O, Al Omari O. Health-Related Stigma, Social Support, Self-Efficacy, and Self-Care Actions Among Adults With Sickle Cell Disease in Oman. Clin Nurs Res. 2022 Jun;31(5):803-811. doi: 10.1177/10547738211046731. Epub 2021 Sep 24. PMID 34555941
- [Background] Castro EM, Van Regenmortel T, Vanhaecht K, Sermeus W, Van Hecke A. Patient empowerment, patient participation and patient-centeredness in hospital care: A concept analysis based on a literature review. Patient Educ Couns. 2016 Dec;99(12):1923-1939. doi: 10.1016/j.pec.2016.07.026. Epub 2016 Jul 18. PMID 27450481
- [Background] Cheng L, Sit JWH, Choi KC, Chair SY, Li X, Wu Y, Long J, Yang H. The effects of an empowerment-based self-management intervention on empowerment level, psychological distress, and quality of life in patients with poorly controlled type 2 diabetes: A randomized controlled trial. Int J Nurs Stud. 2021 Apr;116:103407. doi: 10.1016/j.ijnurstu.2019.103407. Epub 2019 Sep 5. PMID 31679744
- [Background] Crosby LE, Hood A, Kidwell K, Nwankwo C, Peugh J, Strong H, Quinn C, Britto MT. Improving self-management in adolescents with sickle cell disease. Pediatr Blood Cancer. 2020 Oct;67(10):e28492. doi: 10.1002/pbc.28492. Epub 2020 Jul 22. PMID 32697889